CLINICAL TRIAL: NCT00138892
Title: A Randomized Controlled Trial of Long Versus Short Wait For Primary Total Hip and Knee Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: C01-0407; V02-0186
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2011-10-14 (Estimated); Status verified 2011-10

CONDITIONS: Osteoarthritis
Keywords: Quality of life; waiting time; total joint replacement
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Waiting time (access time to Total joint replacement) — See Detailed Description.

SUMMARY:
The primary research question is: Does expedited hip and knee replacement result in improved lower-extremity function at 36 months post randomization as measured by the Western Ontario McMaster Universities Osteoarthritis Index (WOMAC)? A secondary component to this question is whether expedited surgery improves pain and stiffness scores as measured by the WOMAC and generic QOL as measured by the Medical Outcomes Study Short-Form 36 (SF-36) and Health Utilities Index Mark 3 (HUI3)? Secondary questions are: Does joint-specific and generic QOL deteriorate significantly during waiting? Does prolonged waiting increase the economic cost associated with hip and knee arthroplasty? And does expedited surgery have an effect on patient satisfaction with major joint replacement?

DETAILED DESCRIPTION:
Background Long waiting times for certain medical, diagnostic and surgical procedures are the result of high demand for relatively scarce resources. Most western countries have established queues for elective procedures and consultations. Among elective surgical procedures, total hip and knee replacements have the longest waiting lists, twice as long as waits for elective cardiovascular and eye surgery. The data on waiting lists are not highly reliable, nevertheless it is clear that in British Columbia the wait for hip and knee arthroplasty grew from 2 months 1995 to 6 months in 1999 and that a similar increase took place in Ontario. At Vancouver Hospital the median wait for these procedures over the past year has been 7-8 months. Patients are not usually considered candidates for hip or knee replacement until pain and dysfunction have become severe. But waiting prolongs dysfunction and pain that already warrant surgery. A number of studies have demonstrated the burden of suffering that could be relieved by short waits. The question of whether and how much prompt access to surgery could benefit our patients over the long term has attracted very little research. A study we are proposing will for the first time directly address the short- and long-term benefit of expedited surgery with patient-based measures and economic costs, and will do so using valid reliable methods and instruments so that its results can be clearly understood and widely accepted.

Objectives The primary research question is: Does expedited hip and knee replacement result in improved lower-extremity function at 36 months post randomization as measured by the WOMAC functional dimension? A secondary component to the functional question is whether expedited surgery improves pain and stiffness scores as measured by WOMAC and generic quality of life (QOL) as measured by SF-36 and HUI3? Secondary questions are: Does joint-specific and generic QOL deteriorate significantly during waiting? Does prolonged waiting increase the economic cost associated with hip and knee arthroplasty? And does expedited surgery have an effect on patient satisfaction with major joint replacement? Hypothesis Reducing waiting time may improve patient outcomes. This is biologically plausible that prolonging the arthritic process in these joints may result in muscle atrophy, tissue contractures and deterioration of general medical condition that may not be fully recoverable post-surgery. There is some evidence for the harm concurrent with waiting but none for its deleterious long-term effects on hip and knee replacement patients. Our hypothesis is that prolonged waiting is a significant independent risk factor for reduced long-term benefit following surgery. Our secondary hypothesis is that prolonged waiting for hip and knee arthroplasty increases the total economic cost associated with treatment of these disorders.

Research plan The plan involves a randomized controlled clinical trial assigning joint replacement candidates to either a 1-2 month wait or a 7-8 month wait. We will ask patients on both waiting lists to complete QOL and economic assessment questionnaires at the start of waiting, the end of waiting and every six months for 36 months post randomization. Outcome measures will be the WOMAC, the Oxford 12-Item Hip and Knee score, the SF-36, the HUI3, resource utilization information drawn from patient questionnaires and administrative databases, and a measure of patient satisfaction. The analysis will use univariate and multivariate predictive models. In addition we will be assess health trajectories and relative utilization costs.

ELIGIBILITY:
Inclusion Criteria:

All candidates for primary total hip and knee arthroplasty with a diagnosis of osteoarthritis or a¬vascular necrosis. Osteoarthritis is defined by the ACR clinical classification criteria for OA of the hip and knee. , (see Appendix, Table 3, ACR Clinical Classification Criteria). Urgency is not assessed since there are no valid criteria available.

Exclusion Criteria:

(1) Unwillingness to have surgery within 1-2 months, (2) Previous arthroplasty to the index joint, (3) inflammatory arthritis, (4) indications for arthroplasty in >1 joint (any combination of hip or knee, primary or revision) (5) inability to respond to a questionnaire in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2002-08; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
lower-extremity function at 36 months post randomization as measured by the WOMAC functional dimension | 36 months

SECONDARY OUTCOMES:
lower-extremity pain and stiffness at 36 months post randomization as measured by the WOMAC pain and stiffness dimension | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Donald Garbuz, MD, MHSc, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada